CLINICAL TRIAL: NCT04407936
Title: Risk Factors and Prognosis of Adverse Cardiovascular and Kidney Events After Coronary Intervention
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jiyan Chen, Director, Guangdong Provincial People's Hospital
Other Study IDs: GDREC2019555H
Record Dates: First submitted 2020-04-14; First posted 2020-05-29 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Cardio-Renal Syndrome; Coronary Angiography; Coronary Artery Disease; Kidney Diseases; Metabolic Syndrome
Keywords: contrast-induced acute kidney injury; contrast medium; creatinine clearance; coronary angiography; chronic kidney disease; Adverse Cardiovascular and Kidney Events
MeSH Terms: conditions — Cardio-Renal Syndrome; Coronary Artery Disease; Kidney Diseases; Metabolic Syndrome; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- coronary angiography: The investigators recruit all consecutive patients who were undergoing coronary angiography or percutaneous coronary intervention

SUMMARY:
As a single center, retrospective observation study in Guangdong Institute of Cardiovascular Diseases, this study included the main study population of patients who underwent coronary angiography and / or coronary intervention from January 2007 to Decemeber 2018. The hospitalization information was collected in the form of direct derivation of the case, and cardiac and renal adverse events were collected through outpatient recorder system. All-cause death information was obtained from the Public Security and matched to the electronic Clinical Management System of the Guangdong Provincial People's Hospital records.

DETAILED DESCRIPTION:
This is a single center, retrospective observation study collecting data on 88938 coronary angiography and / or coronary intervention patients from January 2007 to Decemeber 2018. Data regarding demographic information, admission diagnoses and history of present illness, biomarkers and details on preventive hydration and medications will be collected. The primary endpoint of this study is All-cause mortality, and secondary endpoints are Adverse Cardiovascular and Kidney Events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to CAG or PCI;

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators reviewed all consecutive patients who were undergoing coronary angiography
Sampling Method: Probability Sample
Enrollment: 88938 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | From hospital admission to 13 years follow-up
  Admission Patients Died for all-cause mortality within 13 years.

SECONDARY OUTCOMES:
Contrast-Induced Acute Kidney Injury (CI-AKI 0.3) | 48 hours
  defined as a ≥ 0.3 mg/dL absolute increase in serum creatinine from baseline during the first 48 hours after the procedure
Cystatin C based CI-AKI (CI-AKI cyc) | 24-48 hours
  Cystatin C based CI-AKI, defined as a ≥10% absolute increase in serum cystatin C during the first 24 hours after the procedure and and a ≥ 0.3 mg/dL absolute increase in serum creatinine from baseline during the first 48 hours after the procedure.mg/dL absolute increase in serum creatinine from baseline during the first 48 hours after the procedure
The change of eGFR, calculate based on CrCl and serum cystatin C | 48-72 hours
  The eGFR creatinine-cystatin C was calculated by the 2012 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) cystatin C equation: 135 *min(Scr/κ, 1)α * max(Scr/κ, 1)-0.601 * min(Scys/0.8, 1)-0.375 * max (Scys/0.8, 1)-0.711 * 0.995Age [* 0.969 if female] [* 1.08 if black], where Scr is serum creatinine, Scys is serum cystatin C, κ is 0.7 for females and 0.9 for males, α is -0.248 for females and -0.207 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1.
Contrast-induced Persistent kidney injury (CI-PKI) | 3 months
  Serum creatinine was measured by endpoint colorimetry or enzymatic assays. CI-PKI was defined as residual impairment of renal function indicated by a ≥ 25% reduction in creatinine clearance at 3 months in comparison with baseline. comparison with baseline
Incidence of major adverse cardiovascular events | 3-12months
  all-cause mortality (cardiovascular and noncardiovascular) and cardiovascular events.
Follow-up major adverse cardiovascular and clinical events | 3-12months
  We will follow up the patients by telephone and outpatient service to know the one year all-cause mortality (cardiovascular and noncardiovascular) and cardiovascular events.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Yong, MD,PhD, Study Director — Guangdong Cardiovascular Institute,Guangdong Provincial People's Hospital; Shiqun Chen, MS, Study Director — Guangdong Cardiovascular Institute,Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen S, Huang Z, Liang Y, Zhao X, Aobuliksimu X, Wang B, He Y, Kang Y, Huang H, Li Q, Yao Y, Lu X, Qian X, Xie X, Liu J, Liu Y. Five-year mortality of heart failure with preserved, mildly reduced, and reduced ejection fraction in a 4880 Chinese cohort. ESC Heart Fail. 2022 Aug;9(4):2336-2347. doi: 10.1002/ehf2.13921. Epub 2022 Apr 18. PMID 35437939
- [Derived] Lai W, Zhao X, Yu S, Mai Z, Zhou Y, Huang Z, Li Q, Huang H, Li H, Wei H, Guo D, Xie Y, Li S, Lu H, Liu J, Chen S, Liu Y. Chronic Kidney Disease Increases Risk of Incident HFrEF Following Percutaneous Coronary Intervention. Front Cardiovasc Med. 2022 Apr 1;9:856602. doi: 10.3389/fcvm.2022.856602. eCollection 2022. PMID 35433884
- [Derived] Huang H, Liu J, Bao K, Huang X, Huang D, Wei H, Remutula N, Tuersun T, Lai W, Li Q, Wang B, He Y, Yang H, Chen S, Chen J, Chen K, Tan N, Wang X, Chen L, Liu Y. Prevalence and Mortality of Moderate or Severe Mitral Regurgitation Among Patients Undergoing Percutaneous Coronary Intervention With or Without Heart Failure: Results From CIN Study With 28,358 Patients. Front Cardiovasc Med. 2022 Mar 3;9:796447. doi: 10.3389/fcvm.2022.796447. eCollection 2022. PMID 35310981
- [Derived] Chen L, Huang Z, Zhao X, Liang J, Lu X, He Y, Kang Y, Xie Y, Liu J, Liu Y, Yang J, Yu W, Deng W, Pan Y, Lu J, Yang Y, Xie X, Qian X, Xu Q, Chen L, Chen K, Chen S. Predictors and Mortality for Worsening Left Ventricular Ejection Fraction in Patients With HFpEF. Front Cardiovasc Med. 2022 Feb 24;9:820178. doi: 10.3389/fcvm.2022.820178. eCollection 2022. PMID 35282383
- [Derived] Liu J, Huang Z, Huang H, He Y, Yu Y, Chen G, Liu L, Wang B, Li Q, Lai W, Xu D, Lu J, Yang Y, Chen L, Chen K, Tan N, Chen J, Chen S, Liu Y. Malnutrition in patients with coronary artery disease: Prevalence and mortality in a 46,485 Chinese cohort study. Nutr Metab Cardiovasc Dis. 2022 May;32(5):1186-1194. doi: 10.1016/j.numecd.2021.12.023. Epub 2022 Jan 6. PMID 35260308
- [Derived] Chen S, Huang Z, Chen L, Zhao X, Kang Y, Lai W, Lu X, Zhou Y, He Y, Huang H, Li Q, Liu J, Liang Y, Dong S, Tan N, Liu Y, Chen J. Does Diabetes Mellitus Increase the Short- and Long-Term Mortality in Patients With Critical Acute Myocardial Infarction? Results From American MIMIC-III and Chinese CIN Cohorts. Front Endocrinol (Lausanne). 2021 Dec 14;12:797049. doi: 10.3389/fendo.2021.797049. eCollection 2021. PMID 34970227
- [Derived] Huang Z, Yang Y, Lu J, Liang J, He Y, Yu Y, Huang H, Li Q, Wang B, Li S, Yan Z, Xu D, Liu Y, Chen K, Huang Z, Ni J, Liu J, Chen L, Chen S. Association of Lipoprotein(a)-Associated Mortality and the Estimated Glomerular Filtration Rate Level in Patients Undergoing Coronary Angiography: A 51,500 Cohort Study. Front Cardiovasc Med. 2021 Nov 17;8:747120. doi: 10.3389/fcvm.2021.747120. eCollection 2021. PMID 34869651
- [Derived] Wang B, Guo Z, Liu J, Li H, Mai Z, Lin F, Ying M, Yu Y, Chen S, Li Q, Huang H, Wei W, Yang Y, Dong S, Zhou Y, Chen J, Tan N, Liu Y. Mild Malnutrition Contributes the Greatest to the Poor Prognosis in Coronary Artery Disease With Well-Controlled Low-Density Lipoprotein Cholesterol Levels: A 4,863 Chinese Cohort Study. Front Nutr. 2021 Sep 29;8:725537. doi: 10.3389/fnut.2021.725537. eCollection 2021. PMID 34660661
- [Derived] Mai Z, Huang Z, Lai W, Li H, Wang B, Huang S, Shi Y, Yu S, Hu Q, Liu J, Zhang L, Liu Y, Chen J, Liang Y, Zhong S, Chen S. Association of Malnutrition, Left Ventricular Ejection Fraction Category, and Mortality in Patients Undergoing Coronary Angiography: A Cohort With 45,826 Patients. Front Nutr. 2021 Sep 16;8:740746. doi: 10.3389/fnut.2021.740746. eCollection 2021. PMID 34604285
- [Derived] Liu J, Li Q, Lai D, Chen G, Wang B, Liu L, Huang H, Lun Z, Ying M, Chen G, Huang Z, Xu D, Meng L, Yan X, Qiu W, Tan N, Chen J, Liu Y, Chen S. Trends in incidence and long-term prognosis of acute kidney injury following coronary angiography in Chinese cohort with 11,943 patients from 2013 to 2017: an observational study. BMC Nephrol. 2021 Jun 25;22(1):235. doi: 10.1186/s12882-021-02427-6. PMID 34172005